CLINICAL TRIAL: NCT07210541
Title: Safety, Clinical Efficacy and Time-to-event Survival in Patients With Degenerative Aortic Valve Disease Scheduled for Stented Biological Aortic Valve Replacement Versus Allograft Aortic Root Replacement.
Brief Title: Comparative Analysis of Stented Biological Prosthesis Versus Aortic Allograft in Patients With Degenerative Aortic Valve Disease
Acronym: BIOCHOICE
Status: Completed | Type: Observational
Sponsor: Chelyabinsk Regional Clinical Hospital (Other Government)
Responsible Party: Principal Investigator, Mikhail Nuzhdin, Director, Chelyabinsk Regional Clinical Hospital
Other Study IDs: 30092025
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-08

CONDITIONS: Bioprosthesis Failure; Allograft
Keywords: aortic valve; bioprosthesis; allograft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stented biological prosthesis: Patients who underwent aortic valve replacement with stented biological valve
  Interventions: Procedure: aortic valve/root replacement
- Allograft aortic root replacement: Patients who underwent allograft aortic root replacement

INTERVENTIONS:
Procedure: aortic valve/root replacement — Aortic valve or aortic root replacement with stented biological prosthesis or aortic allograft
  Groups: Stented biological prosthesis

SUMMARY:
The aim of the observational study is to compare safety, clinical efficacy and time-to-event survival in patients age of 60-74 years with degenerative aortic valve disease that underwent aortic valve replacement with either stented biological prosthesis or aortic allograft.

DETAILED DESCRIPTION:
Early safety included morbidity, mortality rate, freedom from any valve related complications Clinical efficacy included mid-term survival, freedom from reoperation, repeat endocarditis and other valve related complication Time-to-event analysis included freedom from all-cause and cardio-vascular mortality, freedom from stroke, major bleeding, endocarditis, structural valve deterioration and reoperation

ELIGIBILITY:
Inclusion Criteria:

* Patients with degenerative aortic valve disease not emendable for aortic valve repair
* Elective surgery

Exclusion Criteria:

* Left ventricle ejection fraction less than 40%
* Redo surgery
* Indication for concomitant mitral valve replacement
* Aortic valve/root endocarditis
* Severe COPD
* Dialysis patients

Ages: 60 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with degenerative aortic valve disease, age 60-74 years
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2017-01-12 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  Early cardio-vascular mortality

SECONDARY OUTCOMES:
Mortality | 2 years
  Cardio-vascular mortality
Mortality | 2 years
  All-cause mortality
Structural valve deterioration | 2 years
  New onset aortic regurgitation (vc >0,6) or escalated mean pressure gradient over 20 mmHg.
Stroke | 2 years
  Ischemic stroke
Reoperation | 2 years
  Reoperation for valve failure
Endocarditis | 2 years
  Prosthetic valve endocarditis

IPD SHARING:
Plan to Share IPD: No